CLINICAL TRIAL: NCT05113719
Title: Investigation of the Effect of Bridge Exercise Performed at Different Knee Angles on Muscle Strength and Endurance in Healthy Cases
Brief Title: Effect of Bridge Exercise Performed at Different Knee Angles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fettah Saygılı, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Brige Exercise
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: Healthy individuals; Bridge exercise; muscle strenght; core endurance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bridge exercise at knee angle 45 degree (Experimental): The group will perform the bridge exercise at a 45-degree knee flexion angle.
  Interventions: Other: Exercise
- Bridge exercise at knee angle 60 degree (Experimental): The group will perform the bridge exercise at a 60-degree knee flexion angle.
  Interventions: Other: Exercise
- Bridge exercise at knee angle 90 degree (Experimental): The group will perform the bridge exercise at a 90-degree knee flexion angle.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both groups will perform bridge exercise

SUMMARY:
Stabilization exercises help increase strength, stability, balance, gait, and endurance through effective abdominal training. Bridge exercise, which is one of the closed kinetic exercises, is one of the most used spinal stabilization exercises. Although that exercise affects on the trunk muscles, it has been stated that it is related to all muscles of the lower extremity.There are some studies, which are examining the activation of the gluteus maximus, quadriceps, rectus abdominus, iliocostalis lumborum, iliocostalis thoracis, and gastrocnemius muscles while exercising the bridge. Although there are some studies investigating the activation of muscles at different knee angles, there is no study in the literature examining the effect of bridge exercise performed at different knee angles on the strength and endurance of lower extremity and trunk muscles. For these reasons, this study aimed to examine the effect of bridging exercises performed at different knee angles on muscle strength and endurance in healthy subjects.

DETAILED DESCRIPTION:
Participants included in the study will randomly divide into 3 different groups by using simple sealed envelope randomization method. Participants in the first group will perform exercise at knee angle was 45⁰ flexion, the participants in the second group will perform to exercise at knee angle 60⁰ flexion and the participants in the third group will perform exercise knee angle at 90⁰ flexion. All participants will include in a bridging exercise program by a blind researcher at predetermined knee angles (45⁰, 60⁰ 90⁰), 3 sets of 15 repetitions per day, 3 days a week for 6 weeks. Evaluations will be done by a blinded researcher 1 week before starting the 6-week exercise program and 1 week after they finished the program. All evaluations will be made by the same physiotherapist by meeting with participants face to face. Inclusion in the research will be on a voluntary basis. As outcome measures, muscle strength assessment and core Endurance Assessment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-27
* Not having any health problems diagnosed in terms of starting the exercise program
* Individuals who do not exercise regularly

Exclusion Criteria:

* Having any identified health problem that would prevent the exercise
* Individuals who exercise regularly

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Assessment-Baseline | Assessment will be conducted before intervention.
  PowerTrack II Command will be used. The back extensor muscle group and M. Gluteus Maximus, M. Quadriceps Femoris, M. Gastrocinemius muscles of the participants will be evaluated.
Muscle Strength Assessment-Post intervention | Assessment will be conducted immediately after the intervention.
  PowerTrack II Command will be used. The back extensor muscle group and M. Gluteus Maximus, M. Quadriceps Femoris, M. Gastrocinemius muscles of the participants will be evaluated.
Abdominal Muscle Strength Assessment-Baseline | Assessment will be conducted before intervention.
  Manual Muscle Test will be used.
Abdominal Muscle Strength Assessment-Post intervention | Assessment will be conducted immediately after the intervention.
  Manual Muscle Test will be used.
Core Endurance Assessment-1-Baseline | Assessment will be conducted before intervention.
  Prone Plank Endurance Test
Core Endurance Assessment-1-Post intervention | Assessment will be conducted immediately after the intervention.
  Prone Plank Endurance Test
Core Endurance Assessment-2-Baseline | Assessment will be conducted before intervention.
  Squat Endurance Test
Core Endurance Assessment-2-Post intervention | Assessment will be conducted immediately after the intervention.
  Squat Endurance Test
Core Endurance Assessment-3-Baseline | Assessment will be conducted before intervention.
  Dynamic Abdominal Endurance Test
Core Endurance Assessment-3-Post intervention | Assessment will be conducted immediately after the intervention.
  Dynamic Abdominal Endurance Test

CONTACTS AND LOCATIONS:
Overall Officials: Fettah SAYGILI, PT, M.Sc., Study Chair — Research Assistant
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- See also: Related info — https://link.springer.com/article/10.1007/s00586-012-2254-7